CLINICAL TRIAL: NCT02194504
Title: The Belly Fat Study: Nutritional Intervention to Improve Metabolic Health in Subjects With Increased Abdominal Adiposity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NL44614.081.13
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Abdominal Obesity; Liver Fat
Keywords: Metabolic health; Phenotyping; Abdominal obesity; Abdominal adiposity; Liver fat; Belly fat
MeSH Terms: conditions — Obesity, Abdominal; Fatty Liver | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No dietary advice (No Intervention): No dietary intervention
- Dietary advice, Targeted (Experimental): 12-wk dietary advice
  Interventions: Other: Dietary advice, Targeted
- Dietary advice, Western (Experimental): 12-wk dietary advice
  Interventions: Other: Dietary advice, Western

INTERVENTIONS:
Other: Dietary advice, Western — Dietary advice, guided by professional dieticians. Caloric restricted (-30en%) diet with Western type nutrient composition (SFA, carbohydrates, sugars, fruit juice, meat, dairy)
  Arms: Dietary advice, Western
Other: Dietary advice, Targeted — Dietary advice, guided by professional dieticians. Caloric restricted (-30en%) diet with nutrient composition aiming at an improvement in organ health and a reduction in liver fat (PUFA, fish, soy protein, whole grain)
  Arms: Dietary advice, Targeted

SUMMARY:
In the Belly Fat study, the effects of two different caloric-restricted diets on metabolic health will be examined in male and female subjects with increased abdominal adiposity (BMI >27 kg/m2). Metabolic health is defined as health of the primary metabolic organs the liver, gut and the adipose tissue, examined in a static state as well as after the application of a challenge test.

The diets are equally caloric-restricted, but differ in nutrient composition. It is hypothesized that one of the two diets causes a larger improvement in organ health and reduction in liver fat.

DETAILED DESCRIPTION:
Rationale: It is known that in particular visceral fat (abdominal obesity) and fat deposition in non-adipose tissue such as the liver are important factors related to metabolic health, such as the degree of insulin resistance, dyslipidaemia and other well-established cardio-metabolic risk factors. The arise of pathological consequences of abdominal obesity are a result of a disturbance in the elegant interplay between metabolic organs, such as the liver, adipose tissue and gut. Several nutrients have demonstrated to exert positive or negative effects on the health and functioning of metabolic organs. A diet (whole dietary approach) can thus be a power tool to improve the health status of individuals with abdominal obesity by improving organ health.

Objective: The primary objective of this study is to compare the effects of two different diets on the static metabolic health status as assessed by determination of organ health and, more specifically, of lipid accumulation in the liver. The application of a mixed meal challenge test will be used to gain insight in the dynamic metabolic health status. A secondary objective is to determine the reaction (brain activity) of individuals with abdominal obesity after visual and olfactory food-cues.

Study design and intervention: Randomized, parallel design consisting of three groups:

1. 40 subjects, 12-wk nutritional intervention based on dietary advice: diet with 30% caloric restriction and a Western style nutrient composition
2. 40 subjects, 12-wk nutritional intervention based on dietary advice: diet with 30% caloric restriction with a nutrient composition aimed at improving organ health and reducing liver fat
3. 30 subjects, control group, no nutritional intervention (optional: dietary advice at the end of the study period)

Measurements on metabolic health will be conducted at baseline and after 12-wk intervention and include:

* MR imaging for determining body fat distribution
* MR spectroscopy for quantification of liver fat
* Blood sampling (plasma and PBMCs) before and several timepoints after mixed meal challenge
* Adipose tissue sampling before and after mixed meal challenge
* Vascular measurements before and after mixed meal challenge
* Urine and feces sampling

Study population: Males and females, 40-70 yrs old, BMI > 27 kg/m2

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70y at the time of recruitment
* BMI >27kg/m2 or waist circumference >102cm (males) or >88cm (females)

Exclusion Criteria:

* Diabetic (normoglycemic according to WHO criteria (OGTT, fasting blood glucose< 7 mmol/L, after 2 hr <11.1 mmol/L)
* Daily intake of alcohol of >30g (men) or >20g (women)
* Tobacco smoker
* Abuse of drugs
* Any medical conditions or (metal) devices interfering with or posing a risk for the participant in 1H-MRS/MRI scanning (e.g. claustrophobia, pace maker, surgical screws/pins, artificial joints or heart valves, etc.)
* Diagnosed with any long-term medical condition (i.e. cardiovascular disease, gastrointestinal disease, renal dysfunction)
* Use of medications known to interfere with glucose or lipid homeostasis (i.e. corticosteroids)
* Allergic to fish oil or unwilling to consume fish oil supplements
* Unwilling to comply with dietary guidelines
* Restricted to a vegetarian dietary regime

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Intrahepatic lipid accumulation (IHL) | Baseline and after 12-wk intervention
  Assessment of IHL by means of 1H-MRS (magnetic resonance spectroscopy)
Body fat distribution | Baseline and after 12-wk intervention
  Assessment of body fat distribution (SAT/VAT) by means of MRI (magnetic resonance imaging)
Adipose tissue gene expression before and 4h after a mixed meal challenge | Baseline and after 12-wk intervention
  Micro-array/qPCR
Markers of liver health (plasma) before and after mixed meal challenge | Baseline and after 12-wk intervention
  Liver enzymes
Cardio-metabolic risk factors (plasma) before and after mixed meal challenge | Baseline and after 12-wk intervention
  Insulin, glucose, Tg
Inflammatory markers (plasma) before and after mixed meal challenge | Baseline and after 12-wk intervention
  Cytokines
Markers of adipose tissue health (plasma) | Baseline and after 12-wk intervention
  Adipokines
Markers of gut health (plasma) | Baseline and after 12-wk intervention
  Gut hormones
Microbiota (faeces) | Baseline and after 12-wk intervention
Urinary metabolites | Baseline and after 12-wk intervention
PBMC gene expression profile | Baseline and after 12-wk intervention
  Micro-array/qPCR
Vascular functions (blood pressure and arterial stiffness) before and after mixed meal challenge | Baseline and after 12-wk intervention
  PWA

SECONDARY OUTCOMES:
Satiety and wellbeing before and after mixed meal challenge | Baseline and after 12-wk intervention
  Assessment by validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: L Afman, PhD, Principal Investigator — Wageningen University. Department Human Nutrition. Nutrition, Metabolism & Genomics Group

REFERENCES:
- [Derived] Fang Y, Hooiveld GJEJ, Afman LA. Mixed-meal challenge differentially modulates metabolic pathways in adipose tissue in healthy abdominally obese subjects with high versus low liver fat: a secondary analysis of a randomized clinical trial. Nutr Metab (Lond). 2025 Oct 1;22(1):112. doi: 10.1186/s12986-025-01010-2. PMID 41034990
- [Derived] Wang Y, Balvers MGJ, Esser D, Schutte S, Vincken JP, Afman LA, Witkamp RF, Meijerink J. Nutrient composition of different energy-restricted diets determines plasma endocannabinoid profiles and adipose tissue DAGL-alpha expression; a 12-week randomized controlled trial in subjects with abdominal obesity. J Nutr Biochem. 2024 Jun;128:109605. doi: 10.1016/j.jnutbio.2024.109605. Epub 2024 Feb 23. PMID 38401691
- [Derived] Schutte S, Esser D, Siebelink E, Michielsen CJR, Daanje M, Matualatupauw JC, Boshuizen HC, Mensink M, Afman LA; Wageningen Belly Fat Study team. Diverging metabolic effects of 2 energy-restricted diets differing in nutrient quality: a 12-week randomized controlled trial in subjects with abdominal obesity. Am J Clin Nutr. 2022 Jul 6;116(1):132-150. doi: 10.1093/ajcn/nqac025. PMID 35102369